CLINICAL TRIAL: NCT03128905
Title: Colchicine or Prednisone for the Treatment of Acute Calcium Pyrophosphate Deposition (CPPD) Arthritis: Open-label, Randomized, Multicenter, Equivalence Trial of Efficacy and Safety
Brief Title: Trial of Colchicine Versus Prednisone for the Treatment of Acute CPPD Arthritis
Acronym: COLCHICORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other); Hopital Lariboisière (Other); Bichat Hospital (Other); Valenciennes Hospital Centre (Unknown); Armentières Hospital Centre (Unknown); Dunkerque Hospital Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-P0050
Record Dates: First submitted 2017-04-06; First posted 2017-04-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chondrocalcinosis
Keywords: Colchicine; Corticoids; Prednisone; CPPD; Calcium Pyrophosphate Deposition Disease
MeSH Terms: conditions — Chondrocalcinosis

STUDY DESIGN:
Masking Description: No masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Active Comparator): Patients assigned to this group will receive the Colchicine opocalcium 1mg treatment.
  Interventions: Drug: Colchicine opocalcium 1mg
- Prednisone (corticoids) (Experimental): Patients assigned to this group will receive Prednisone : Cortancyl 20mg.
  Interventions: Drug: Prednisone : Cortancyl 20mg

INTERVENTIONS:
Drug: Colchicine opocalcium 1mg — International non-proprietary name: Colchicine
  Molecule owner: Mayoly-Spindler Laboratory, 1mg scored tablet for oral administration, authorized 03/02/1995.
  Composition :
  Active principle : Crystallized colchicine Excipients: Erythrosine aluminium lake, lactose, saccharose, magnesium stearate and povidone.
  Other Names: Mayoly-Spindler laboratory
  Arms: Colchicine
Drug: Prednisone : Cortancyl 20mg — International non-proprietary name: Prednisone
  Molecule owner : SANOFI AVENTIS France 20 mg scored tablet for oral administration, authorized since 02/05/1990, generic drug available.
  Composition :
  Active principle : Prednisone Excipients: Maize starch, lactose, talc, magnesium stearate.
  Other Names: Sanofi Aventis France
  Arms: Prednisone (corticoids)

SUMMARY:
Chondrocalcinosis, recently renamed the calcium pyrophosphate deposition (CPPD) disease, is a very frequent affection of the elderly and causes very painful arthritis.

International recommendations for the treatment of patients suffering from CPPD are based upon rare studies, not randomized, with small samples, and thus very weak scientific evidence.

The treatment of CPPD arthritis is extrapolated from the experience of gout treatment, another crystal deposition disease.

Among recommended treatments, colchicine and oral steroids are recommended as first-line treatments, while NSAIDs are used with caution in elderly populations of patients.

Colchicine utilization is not risk-free, in particular with old patients and patients with renal impairment.

Drug interactions of colchicine can have serious consequences, especially in a polymedicated old patient's population.

Oral steroids are an interesting alternative in this indication with a potential of being better tolerated, but comparative efficacy with colchicine needs to be studied.

From a broader point of view, colchicine and oral steroids have never been compared in any crystal related arthritis.

This is the first large randomized controlled trial for CPPD acute arthritis.

DETAILED DESCRIPTION:
Chondrocalcinosis, recently renamed the calcium pyrophosphate deposition (CPPD) disease, is a very frequent affection of the elderly and causes very painful arthritis.

International recommendations for the treatment of patients suffering from CPPD are based upon rare studies, not randomized, with small samples, and thus very weak scientific evidence.

Some factors are known to trigger CPPD arthritis (trauma, surgery, infection, hospitalization). Prevalence increases with age, and case series estimate the presence of chondrocalcinosis in over 20% of 80 plus years population.

International recommendations for the treatment of patients suffering from CPPD are based upon rare studies, not randomized, with small samples, and thus very weak scientific evidence.

The treatment of CPPD arthritis is extrapolated from the experience of gout treatment, another crystal deposition disease (this one related to monosodium urate crystals that deposit after long-standing hyperuricemia.

Among recommended treatments, colchicine and oral steroids are recommended as first-line treatments, while NSAIDs are used with caution in elderly populations of patients.

Colchicine utilization is not risk-free, in particular with old patients and patients with renal impairment. Drug interactions of colchicine can have serious consequences, especially in a polymedicated old patient's population. Oral steroids offer an interesting alternative with the potential of being better tolerated.

However, even oral steroids are recommended, their efficacy in CPPD arthritis isn't demonstrated. Interesting comparative results with NSAIDs were shown for the treatment of gout flares. These results may not be fully extrapolated to CPPD which holds differences with gout. In addition, oral steroids were not compared to colchicine which is the benchmark treatment in many countries for CPPD.

The aim of this study is to compare the efficacy of colchicine and oral steroids for the treatment of CPPD acute arthritis and compare their tolerance profile. It is the first large randomized controlled trial comparing two treatments of CPPD acute arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 and older
* Patient with mono/polyarticular CPPD acute arthritis
* Hospitalized patient (without infectious syndrome considered insufficiently controlled by the clinicians and diabetic decompensation)
* Diagnosis confirmed :
* By the evidence of CPP crystals on synovial fluid examination.
* By the existence of a typical clinical arthritis (joint pain, erythema, swelling, maximal intensity in less than 24h) AND presence of chondrocalcinosis signs in knee, wrists, or pubic symphysis on plain X-rays or crowned tooth in cervical rachis scan.
* Pain VAS ≥ 40/100 at the enrollment
* Duration of symptoms evolution for less than 36h.
* No prior intake of oral steroids, colchicine or NSAIDs for this acute arthritis.
* Signed patient's consent.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Contraindication to colchicine (creatinine clearance below 30ml/min, severe hepatic dysfunction, macrolide or ongoing pristinamycin or macrolid treatment, …) or corticoids utilization (uncontrolled diabetes, uncontrolled progressive infection, uncontrolled arterial hypertension…)
* Severe cognitive disorders that does not allow patient to evaluate his pain.
* Patient under guardianship, curatorship
* Patient receiving morphinic analgesia.
* Gout history or presence of monosodium urate crystals at the examination of the synovial fluid.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the pain VAS at 24 hours | From the first treatment administration to 24 hours after.
  Evolution of the pain Visual Analog Scale (VAS), between baseline and 24 hours after the first treatment administration, without any recourse to other anti-inflammatory treatments.

SECONDARY OUTCOMES:
Proportion of patients with at least one adverse event within 48 hours | 48 hours following the first administration
  Proportion of patients with at least one adverse event within 48 hours following the first drug intake (diarrhea, abdominal pain, nausea, vomiting, a 50% fasting blood glucose increase, excitability, sleep disorders, high blood pressure apparition [above 140/90mmHg], change in creatinine clearance)
Change from baseline of biological inflammatory syndrome at 48 hours | From the first treatment administration to 48 hours after.
  C Reactive Protein change from baseline 48 hours after the first treatment intake.
Number of joints affected and their localizations | Before, 24 hours and 48 hours after the first administration
  Number of affected articulations and their localization before the first intake, after 24 hours and after 48 hours.
Need of emergency morphinic treatment | 24 hours after the first administration
  Proportion of patients requiring analgesia with morphine within the first 24 hours.
Analgesic consumption | From 24 hours to 48 hours after the first treatment administration
  Proportion of patients requiring additional analgesics between the 24th and 48th hour following the 1st intake.
Proportion of patients with an efficacy response of at least 50% | 24 hours and 48 hours after the first administration.
  Proportion of patients with at least a 50% decrease in pain VAS at 24 and 48 hours after the first intake.
Proportion of patients with an efficacy response of at least 20% | 8, 12 and 24 hours after the first administration.
  Proportion of patients with at least a 20% decrease in pain VAS at 8, 12 and 24 hours after the first administration.
Complete crisis resolution within 7 days | 7 days after 1st administration
  Proportion of patient with a complete resolution of the arthritis within the 7 days after 1st intake (defined by a ≤3/10 VAS score)
Initial crisis resolution delay | 7 days after 1st administration
  Delay to the complete resolution of the arthritis from the first drug intake
Absence of crisis recidivism within 7 days | Within the 7 days following the 1st administration
  Relapse rate within the 7 days following the 1st intake (defined by the recurrence of pain with a >3/10 VAS score)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Houvenagel, Pr, Principal Investigator — Lille Catholic University; Tristan Pascart, Dr, Study Chair — Lille Catholic University
Locations (7):
- France (7):
  - CHRU Lille, Lille, Hauts-de-France
  - Lille Catholic Hospital, Lille, Hauts-de-France
  - CH Valenciennes, Valenciennes, Hauts-de-France
  - Dr Nicolas SEGAUD, Armentières
  - Dr Rémi LEROY, Dunkirk
  - Hôpital de Lariboisière, Paris, Île-de-France Region
  - Hôpital Bichat, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pascart T, Robinet P, Ottaviani S, Leroy R, Segaud N, Pacaud A, Grandjean A, Luraschi H, Rabin T, Deplanque X, Maciejasz P, Visade F, Mackowiak A, Baclet N, Marechaux S, Lefebvre A, Budzik JF, Bardin T, Richette P, Norberciak L, Ducoulombier V, Houvenagel E. Evaluating the safety and short-term equivalence of colchicine versus prednisone in older patients with acute calcium pyrophosphate crystal arthritis (COLCHICORT): an open-label, multicentre, randomised trial. Lancet Rheumatol. 2023 Sep;5(9):e523-e531. doi: 10.1016/S2665-9913(23)00165-0. Epub 2023 Aug 8. PMID 38251496